CLINICAL TRIAL: NCT07088809
Title: Comparative Study Between Hydroxyapetite Nanoparticles and Tricalcium Phosphate Nanoparticles Loaded on Platelet Rich Fibrin Membranes for Treatment of Gingival Recession
Brief Title: Hydroxyapetite Nanoparticles and Tricalcium Phosphate Nanoparticles Loaded on Platelet Rich Fibrin Membranes for Treatment of Gingival Recession
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Enas Elgendy (Other)
Responsible Party: Sponsor-Investigator, Enas Elgendy, Prof of Oral Medicine and Periodontology, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kafrelsheikh 2
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Periodontal Diseases; Gingival Recession Localized Moderate; Nano-hydroxyapatite; Nano Tricalcium Phosphate; Platelet Rich Fibrin
Keywords: gingival recession; nano tricalcium phosphate; nanocrystalline hydroxyapatite; platelet rich plasma
MeSH Terms: conditions — Periodontal Diseases; Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap (Experimental): Ten sites with gingival recession treated with Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap.
  Interventions: Procedure: Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap
- Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap (Experimental): Ten sites of gingival recession treated with Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap
  Interventions: Procedure: Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap

INTERVENTIONS:
Procedure: Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap — Two horizontal incisions were made at right angles to the adjacent interdental papillae at the CEJ level without interfering with the gingival margin of the neighbouring teeth. To mobilize the flap, two oblique vertical releasing incisions were extended beyond the mucogingival junction. A full thick¬ness trapezoidal flap was then elevated up to the mucogingival junction, and follow¬ing penetration of the periosteum, a par¬tial thickness flap was dissected further apically. The papillae mesial and distal to the recession defects were deepithelialized.
  Following conditioning, the root surface was rinsed with sterile saline for 1 minute. Following conditioning, the root surface the PRF membrane loaded by nanocrystale hydroxyapatite was positioned to cover the recession up to CEJ. The flap was then coronally advanced to cover the membrane, and flap was closed using simple interrupted sutures. A periodontal dressing was placed over the recipient site for 10 days to protect the wounds.
  Arms: Nanocrystalline hydroxyapatite loaded in PRF+ coronally advanced flap
Procedure: Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap — Two horizontal incisions were made at right angles to the adjacent interdental papillae at the CEJ level without interfering with the gingival margin of the neighbouring teeth. To mobilize the flap, two oblique vertical releasing incisions were extended beyond the mucogingival junction. A full thick¬ness trapezoidal flap was then elevated up to the mucogingival junction, and follow¬ing penetration of the periosteum, a par¬tial thickness flap was dissected further apically. The papillae mesial and distal to the recession defects were deepithelialized.
  Following conditioning, the root surface was rinsed with sterile saline for 1 minute. Following conditioning, the root surface the PRF membrane loaded by Nanocrystalline tricalcium was positioned to cover the recession up to CEJ. The flap was then coronally advanced to cover the membrane, and flap was closed using simple interrupted sutures. A periodontal dressing was placed over the recipient site for 10 days to protect the wounds.
  Arms: Nanocrystalline tricalcium phosphate (NcTCP) loaded in PRF+ coronally advanced flap

SUMMARY:
The "Glossary of the American of Periodontology" defines gingival recession (GR) as the apical movement of the gingival margin beyond the cement-enamel junction. Therefore, root surface exposure brought on by gingival recession results in cosmetic impairment, fear of tooth loss, increased susceptibility to root caries, and dentin hypersensitivity. The use of free gingival grafts, sliding pedicle grafts, subepithelial connective tissue grafts, envelope or tunnelling techniques, the use of acellular dermal, connective tissue allografts, guided tissue regeneration, and coronally advanced flap (CAF) are the surgical methods that have been developed to treat gingival recession. The medical area has been invaded by nanotechnology, and the findings are highly promising. Nanomaterials perform far better than conventional materials thanks to their superior surface, size, and quantum effects. Hydroxyapatites (HAs) are a family of materials used for bone grafting that have a high level of biocompatibility, which is partly due to their inclusion in naturally calcified tissue. The aim of the present study was to compare between nanocrystalline hydroxyapatite and tricalcium phosphate carried on PRP membrane in treatment of Miller's class 1 gingival recession in human.

DETAILED DESCRIPTION:
The primary objective of periodontal therapy is the regeneration of periodontal tissues that have been lost owing to periodontal disease since gingival recession results in the loss of both soft and hard tissue. Periodontal regeneration, demonstrated histologically by the development of new cementum, new alveolar bone, functionally orientated periodontal ligament, and gingiva, is the rebuilding of the lost tissues. Platelet rich fibrin (PRF), which contains significant amounts of growth factors, platelets, fibrin membrane, leukocytes, and cytokines, was introduced for periodontal regeneration. The capacity of PRF to boost collagen production and fibroblast proliferation has been demonstrated, and it is widely used to repair and enhance the regeneration of both soft tissues and hard tissues following various periodontal surgical procedures. Xenografts were established in the field of periodontology to address the drawbacks of autogenous bone graft and allograft. Although these materials provide a solution to some of the aforementioned issues, the issue of immunogenicity and the transmission of disease had been frequently brought up; as a result, alloplastic materials were produced. These substances, which are artificial, inorganic, and biocompatible bone graft alternatives, offer a potential substitute for the treatment of periodontal disorders. The benefits of these materials include better accessibility, the removal of the requirement for a donor site, and the absence of any risk of disease transmission. In controlled clinical studies, hydroxyapatite (HA) and tricalcium phosphate (TCP), two alloplastic materials, significantly improved clinical outcomes at grafted locations compared to non-grafted sites. Cone beam computed tomography produces 3D images that are required in periodontics for the diagnosis of intra bony defects, furcation involvements, and destructions of the buccal and lingual bones. The objective of this study was to compare the effectiveness of nanocrystalline hydroxyapatite and tricalcium phosphate, both applied on a PRP membrane, in treating Miller's class 1 gingival recession in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good systemic health and no contraindication for periodontal surgery.
* Patients who are able to maintain good oral hygiene.
* Gingival thickness for the site selected should be ≥1mm.
* The height of keratinized gingiva (HKG) for the site selected should be ≥1 mm (HKG is the distance between the most apical point of the gingival margin and the mucogingival junction).

Exclusion Criteria:

* Active infectious diseases (hepatitis, tuberculosis, HIV, etc….).
* Medically compromised patients.
* Patients taking medications known to cause gingival enlargement.
* Pregnant patients and smokers.
* Previous mucogingival surgery at the defect.
* Restorations or caries in the area to be treated and non vital tooth.
* Teeth which are tilted or rotated.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of root coverage (RC) | after 1, 3, 6 months post operatively
  Percentage of root coverage (RC): is calculated after 1, 3, 6 months as [RH preoperative - RH postoperative]/RH preoperative) x 100%.
Facial bone level | 6 months
  Facial bone level was the distance from the apex of the tooth to most coronal point of the facial bone.
Horizontal facial bone thickness | after 6 months
  Horizontal facial bone thickness was the thickness of the facial bone at the middle of the root length.
Recession height (RH) | at 1, 3 and 6 month post surgically
  distance between cemento-enamel junction (CEJ) to the most apical point of the gingival margin (GM).
Recession width (RW) | at 1, 3 and 6 month post surgically
  from one border of the recession to another, measured at the CEJ.
Height of the keratinized tissue (HKT) | 1, 3 and 6 month post surgically
  Height of the keratinized tissue (HKT): distance between the most apical point of the GM and the mucogingival junction (MGJ).

SECONDARY OUTCOMES:
Bone density | after 6 months
  Bone density: measured at the facial bone at the middle of the root length
Plaque index | at 1, 3 and 6 month post surgically
Gingival index (GI) | at 1, 3 and 6 month post surgically
Probing pocket depth (PPD) | at 6 months post surgically
Clinical attachment level (CAL) | at 6 months post surgically
Wound healing index (WHI) | at 14 days and 1, 3, and 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Enas Elgendy, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF